CLINICAL TRIAL: NCT04855149
Title: Satisfaction Survey After Distal Surgery Performed Under Local Infiltration (Walant) or Under Axillary Block
Acronym: WALAX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2020/PC-01
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-04

CONDITIONS: Anesthesiology; Satisfaction, Patient; Surgery
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WALANT: anesthesia performed with WALANT technique
  Interventions: Other: Patient satisfaction
- BAx: anesthesia performed with axillary block under ultrasound control
  Interventions: Other: Patient satisfaction

INTERVENTIONS:
Other: Patient satisfaction — Patient satisfaction evaluated with EVAN LR questionnaire

SUMMARY:
In the 1970s-1980s, Dr. Donald Lalonde (surgeon, Canada) developed an anesthetic technique for hand surgery called WALANT (Wide Awake Local Anesthesia No Tourniquet). This technique is based on the joint administration of a local anesthetic (lidocaine) and epinephrine (adrenaline), which limits bleeding and makes it possible to dispense with a tourniquet. In addition, and contrary to truncal anesthesia, this combination of drugs infiltrated opposite the surgical site preserves the mobility of the limb. However, this technique is not without risk and some adverses events have been reported: intoxication by local anesthetics due to overdose and digital necrosis with the use of procaine or cocaine.

Currently in France, truncal anesthesia with a pneumatic tourniquet on the arm is often preferred for hand surgery (axillary block or BAx). In this case, the pneumatic tourniquet is used to minimize intraoperative blood loss and improve the visibility of the operating field. However, it can be a source of discomfort, pain, or transient neurological deficit.

To date, few studies comparing WALANT and BAx are available and none have evaluated the perioperative experience of patients and the incidence of paresthesias in the short and long term.

In order to measure the perioperative satisfaction of patients undergoing hand surgery with BAx or WALANT, we conduct a prospective observational non-randomized study evaluating the EVAN-LR satisfaction score at D0. The secondary objectives of the study are to evaluate postoperative adverse events (digital necrosis, paresthesias, local anesthetic intoxications, infection of the operated limb), consumption of postoperative analgesic treatments in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yars
* scheduled surgery of the hand, wrist or elbow under local or loco-regional anesthesia
* Consent to participate

Exclusion Criteria:

* contraindication to loco-regional or local anesthesia
* allergy to the products administered (lidocaine, epinephrine)
* pregnant woman
* comprehension disorder (confusion, cognitive disorder...) or linguistic disorder that does not allow answering the follow-up questionnaires
* refusal to participate or to follow up
* surgery in emergency or under general anesthesia

Translated with www.DeepL.com/Translator (free version)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are patients at least 18 years old, hospitalized for scheduled surgery, who have accepted the principle of the study, are able to complete the EVAN-G questionnaire and are able to walk alone.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction of day case surgery | Day 0
  Satisfaction of day case surgery measured with EVAN LR score (EVAN LR : Evaluation du Vécu de l'Anesthésie LocoRégionale; the EVAN-LR comprises 19 items, structured in a global index and five dimensions: Attention, Information, Discomfort, Waiting, and Pain; , All dimensions are scored on a scale from 0 to 100, with 100 indicating the best possible level of satisfaction and 0 the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Principal Investigator — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France